CLINICAL TRIAL: NCT01919931
Title: Immunological and Molecular Interaction Between the Host and Candida Albicans Biofilm
Brief Title: Immunological Interaction Between the Host and Candida Albicans Biofilm
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S55012
Record Dates: First submitted 2013-06-19; First posted 2013-08-09 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Candidiasis
Keywords: Candida albicans; Candidiasis; Biofilm; Flow cytometry; Mannose Binding Lectin
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Samples to be retained: whole blood, Plasma and White cells.

GROUPS / COHORTS (2):
- Candida Infection: Patients infected with Candida albicans
- No infection: Patients with no Candida albicans infection

SUMMARY:
Candida albicans is one of the most common nosocomial infection and the onset relies on the host immune status. The purpose of this study is to determine the immunological profile of patients infected with Candida albicans, that could ideally lead to a strategy to identify patients who could benefit from prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with Candida albicans
* Patients not infected with Candida albicans

Exclusion Criteria:

* Underage patients
* Non consenting patients
* Unconscious patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Candida albicans infection. Patients with no Candida albicans infection. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Immunological phenotyping of patients | 2 months

SECONDARY OUTCOMES:
Mannose Binding Lectin levels | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Liston, Group Leader, Study Director — Flemish Institute of Biotechnology
Locations (1):
- Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant, Belgium